CLINICAL TRIAL: NCT06914024
Title: Clinical Association Between Celiac Disease and Intussusception in Children Attending Assiut University Children Hospital
Brief Title: Clinical Association Between Celiac Disease and Intussusception in Children
Acronym: Celiac
Status: Not yet recruiting | Type: Observational
Sponsor: merna hamdy kamal mohammed (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, merna hamdy kamal mohammed, resident physician, Assiut University
Organization: Assiut University (Other)
Other Study IDs: celiac and intussusception
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Celiac Disease in Children; Intussusception
Keywords: pediatric gastrointestinal disease
MeSH Terms: conditions — Intussusception

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical association Between Celiac Disease and Intussusception in children

ELIGIBILITY:
Inclusion Criteria:

Children aged 6 months to 18 years Diagnosed with celiac disease based on serology and biopsy Diagnosed with intussusception confirmed by imaging Parent or legal guardian provides informed consent

Exclusion Criteria:

Children with known gastrointestinal abnormalities other than celiac disease History of abdominal surgery Incomplete or unavailable medical records Patients on immunosuppressive therapy

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 1. To explore the potential association between celiac disease and intussusception in pediatric patients, identifying any common clinical features or patterns that may suggest a link between the two conditions.
  2. To determine the prevalence of Celiac Disease among children diagnosed with intussusception attending assiut university children hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Celiac Disease and Intussusception | 1year
  Celiac Disease and Intussusception in children

SECONDARY OUTCOMES:
Analysis of clinical characteristics associated with intussusception | 1year
  Analysis of clinical characteristics associated with intussusception in children with celiac disease